CLINICAL TRIAL: NCT00494858
Title: Treatment of Bulimia Nervosa: Dysregulated Subtype
Brief Title: Focused Versus Enhanced Cognitive Behavioral Therapy for Treating Women With Bulimia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH071641 (NIH); K23MH071641 (NIH); DATR AK-TNAI2
Record Dates: First submitted 2007-06-28; First posted 2007-07-02 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Eating Disorders
Keywords: Bulimia nervosa; Cognitive Behavioral Therapy; Personality Disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Personality Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT-EF (Active Comparator): Participants will receive cognitive behavioral therapy - focused
  Interventions: Behavioral: Cognitive behavioral therapy - focused (CBT-EF)
- CBT-EB (Experimental): Participants will receive cognitive behavioral therapy - broad
  Interventions: Behavioral: Cognitive behavioral therapy - broad (EB)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy - focused (CBT-EF) — Focused CBT concentrates only on BN symptoms. There will be 20 sessions over the course of 5 months.
  Arms: CBT-EF
Behavioral: Cognitive behavioral therapy - broad (EB) — Broad CBT addresses symptoms of BN, as well as those of the personality disorder. CBT-EB incorporates ED interventions from CBT-EF but also has modules focused on addressing mood intolerance and interpersonal difficulties. There will be 20 sessions over 5 months.
  Arms: CBT-EB

SUMMARY:
This study will compare the effectiveness of two types of cognitive behavioral therapy in treating adult women with the dysregulated subtype of bulimia nervosa.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a common eating disorder that is characterized by periods of bingeing and purging. People with the dysregulated subtype of BN experience behavioral impulsivity; disruption of cognitive, affective, behavioral, and neurophysiological processes (dysregulation); interpersonal dysfunction; and poor treatment response. To date, no therapies have been tested for this specific population, and it is unknown whether therapy that directly focuses on treating BN symptoms or one that addresses both eating and personality disorder symptoms is more effective. Cognitive behavioral therapy (CBT), which concentrates on modifying patients' behaviors and ways of thinking, has been effective in treating BN. This study will compare the effectiveness of two types of CBT, focused and broad, in treating adult women with the dysregulated subtype of BN.

Participants in this single-blind study will be randomly assigned to receive 20 sessions of either broad (enhanced) or focused CBT. Participants will meet with a therapist once or twice weekly until 20 sessions have occurred. Broad CBT will address symptoms of BN, as well as those of the personality disorder. Focused CBT will concentrate only on BN symptoms. Before treatment begins, participants will complete a set of questionnaires pertaining to their experiences with BN, depression, anxiety, and interpersonal relationships. The questionnaires will be used throughout the study to assess participants' progress. Participants will also attend a clinical interview lasting approximately 3.5 hours. Questions will concern BN, other eating disorder symptoms, depression, anxiety, and interpersonal relationships. Blood samples and vital signs will also be taken at the time of the clinical interview and as needed later in the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bulimia nervosa
* Presence of borderline personality disorder features
* History of one mood or anxiety episode within 2 years prior to study entry
* If taking psychiatric medication, dose has been stable for at least 6 weeks at time of study entry

Exclusion Criteria:

* Substance dependence
* Diagnosis of bipolar I disorder
* Psychosis
* Mental retardation
* Receiving psychosocial treatment

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms | Measured throughout the study

SECONDARY OUTCOMES:
Depression symptoms | Measured throughout the study
Anxiety symptoms | Measured throughout the study
Interpersonal relationships | Measured throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Heather Thompson-Brenner, PhD, Principal Investigator — Center for Anxiety and Related Disorders, Boston University
Locations (1):
- Center for Anxiety and Related Disorders, Boston University, Boston, Massachusetts, United States